CLINICAL TRIAL: NCT00643188
Title: Catheter Ablation Versus Standard Conventional Treatment in Patients With Left Ventricular Dysfunction and Atrial Fibrillation
Brief Title: Catheter Ablation vs. Standard Conventional Treatment in Patients With LV Dysfunction and AF
Acronym: CASTLE-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP020
Record Dates: First submitted 2008-02-22; First posted 2008-03-26 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Atrial fibrillation; Ablation; Heart failure; Home Monitoring
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Radiofrequency ablation of atrial fibrillation:
  Subjects assigned to the catheter AF ablation strategy will undergo ablation within 48 hours after baseline evaluation. The aim of the procedure is to achieve isolation of all Pulmonary Veins (PVs) and to restore sinus rhythm. Only radiofrequency catheter based AF ablation is permitted; other methods, like cryoablation, ultrasound and laser, are not permitted in this study.
  Before ablation, a transesophageal echocardiogram must be performed in order to rule out presence of atrial thrombi.
  Anticoagulation should be initiated, or continued, for at least six months post ablation. Six months after successful ablation and in absence of any recurrence of AF, antiarrhythmic drugs should be discontinued.
  Interventions: Procedure: Radiofrequency ablation
- 2 (Active Comparator): Conventional treatment:
  Subjects assigned to the conventional treatment strategy will be treated according to current guidelines for the management of patients with chronic heart failure and/or atrial fibrillation. Efforts to maintain sinus rhythm in this study arm are recommended.
  Anticoagulation will be initiated, if not already started, and maintained throughout the study according to current guidelines.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation of atrial fibrillation
  Arms: 1
Other: Conventional treatment — The best medical treatment according to the ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult and the ACC/AHA/ESC 2006 Guidelines for Management of Patients with Atrial Fibrillation.
  Arms: 2

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice. The incidence and prevalence of AF increase exponentially with increasing age and AF is associated with higher mortality, more frequent hospitalization, and lower quality of life. Furthermore, AF is often associated with heart failure. The majority of AF is initiated by ectopic foci found primarily in the pulmonary veins. It was shown that catheter ablation of those veins could eliminate episodes of AF. In patients with heart failure, catheter ablation could improve cardiac function, symptoms and quality of life. It remains still unknown whether AF ablation is more effective than conventional treatment in terms of mortality and morbidity.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice; its incidence and prevalence increase exponentially with increasing age and it is associated with increased mortality, more frequent hospitalization, and decreased quality of life.

An initial approach to the cure of patients suffering from AF was surgical intervention with the Maze procedure, which involved the creation of linear lesions in the atria to break the re-entrant wavefronts responsible for maintenance of AF. Subsequently, less invasive procedures have been developed to achieve the same results. One of them is catheter based radio frequency ablation, in which a catheter is placed in the heart percutaneously, followed by application of electrical energy to the target regions, thereby creating a permanent lesion.

The origin of AF is often localized in the pulmonary veins (PVs); therefore one common approach is to ablate them in order to electrically isolate them from the left atrium (LA). Several strategies have been developed, such as linear, segmental, circumferential, and double-lasso.

Additionally, other anatomical regions such as the right atrium (RA), superior vena cava (SVC), and coronary sinus (CS) can be ablated in order to eliminate non-PV drivers of AF.

Heart failure (HF) is frequently a chronic and lethal condition, causing substantial morbidity and, after initial diagnosis, results in mortality rates which come close to or exceed those of many malignancies.

Both AF and HF have a significant impact on the health care expenditures. The two diseases often coexist, there is a complex interaction between them: many of the processes that predispose to HF, such as hypertension, diabetes, coronary artery disease, and valvular heart disease, are also risk factors for the development of AF. Similarly, many of the echocardiographic findings that are common in patients with HF, including LA enlargement, increased left ventricular (LV) wall thickness, and reduced LV fractional shortening, predispose patients in the development of AF.

In small groups of patients suffering from HF and AF, radio frequency ablation has been performed; the restoration of sinus rhythm resulted in the improvement of quality of life, exercise performance, and cardiac parameters like ejection fraction and fractional shortening. It is still unknown if such therapy is also effective in reducing mortality and morbidity.

CASTLE-AF is a prospective, unblinded, randomized, multicenter study whose aim is to compare the effect of radio frequency catheter-based ablation on mortality and morbidity with that of conventional treatment in HF subjects with AF. About 420 patients with LV dysfunction (ejection fraction ≤ 35%) and New York Heart Association (NYHA) class ≥ II, already implanted with a dual chamber implantable cardioverter defibrillator (ICD) with Home Monitoring® capabilities, will be enrolled and randomized 1:1 to undergo either AF ablation or standard treatment as indicated in the American College of Cardiology (ACC)/American Heart Association (AHA)/European Society of Cardiology (ESC) 2006 guidelines for the management of patients with AF. In addition to planned and unplanned visits, the ablated patients will be constantly monitored remotely via Home Monitoring®, in order to detect any recurrences of AF episodes, even if non-symptomatic or short in duration, during an observational period of minimum 3 years for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal or persistent atrial fibrillation
* Failure or intolerance of antiarrhythmic drug therapy or unwillingness to take antiarrhythmic drugs
* Left Ventricular Ejection Fraction <= 35%
* NYHA >= II
* ICD for primary or secondary prevention with atrial sensing capabilities or Cardiac Resynchronization Therapy plus Defibrillator (CRT-D) device, both with Home Monitoring® technology already implanted
* Patient is willing and able to comply with the protocol and has written informed consent
* Age >= 18 years

Exclusion Criteria:

* Contraindication for chronic anticoagulation therapy and heparin
* Documented left atrial diameter > 6 cm
* Previous left heart ablation procedure for atrial fibrillation
* Acute coronary syndrome, cardiac surgery, angioplasty or stroke within 2 months prior to enrollment
* Untreated hypothyroidism or hyperthyroidism
* Enrollment in another investigational drug or device study
* Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertility age
* Mental or physical inability to take part in the study
* Listed for heart transplant
* Cardiac assist device implanted
* Planned cardiovascular intervention
* Life expectancy ≤ 12 months
* Uncontrolled hypertension
* Requirement for dialysis due to terminal renal failure
* Participation in another telemonitoring concept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
All-cause mortality or worsening heart failure requiring unplanned hospitalization | 7 years

SECONDARY OUTCOMES:
All-cause mortality Cardiovascular mortality Unplanned hospitalization due to cardiovascular reason Worsening heart failure requiring unplanned hospitalization Cerebrovascular accidents Left ventricular function Exercise tolerance Quality of life | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Brachmann, Prof. Dr., Study Chair — Klinikum Coburg, Germany; Nassir F. Marrouche, Dr., Study Chair — Division of Cardiology, University of Utah Health Sciences Cente, Salt Lake City, Utah, United States
Locations (32):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide
  - Royal Brisbane and Women's Hospital, Herston
- Austria (2):
  - A. ö. Krankenhaus der Elisabethinen Linz, Linz
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Germany (17):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Charité Campus Mitte, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Franz-Volhard-Klinik, Universitätsklinikum Charité, Berlin
  - Vivantes-Klinikum am Urban, Berlin
  - Städtische Kliniken Bielefeld, Bielefeld
  - St. Marien Hospital, Bonn
  - Zentralkrankenhaus Links der Weser, Siebels & Langes Partnerschaft, Bremen
  - Klinikum Coburg, Coburg
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Kardiocentrum Frankfurt an der Klinik Rotes Kreuz, Frankfurt am Main
  - Universitätsklinikum der Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Krankenhaus Landshut-Achdorf, Landshut
  - Klinikum Lüdenscheid, Lüdenscheid
  - Deutsches Herzzentrum München, München
  - St. Vincenz-Krankenhaus, Paderborn
  - Universitätsklinikum Rostock, Rostock
- Hungary (2):
  - Semmelweis Medical University, Budapest
  - The Debrecen University of Medicine, Debrecen
- Netherlands (3):
  - Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Isala Klinieken, Zwolle
- National Institute of Cardiology, Warsaw, Poland
- Russia (4):
  - HRD Surgical Department; Federal Centre of Cardiovascular Surgery, Krasnoyarsk
  - N.S.B.R.I. of Circulation Pathology, Novosibirsk
  - Arrhythmology Department; Federal Heart Blood and Endocrinology Center n.a. V. A. Almazov, Saint Petersburg
  - FSBI Research Institute of Cardiology, Siberian Branch of RAMS, Tomsk
- The Heart Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to publish results of this investigation in peer-reviewed journals (online: open-access), but it is not yet decided to annex individual participant data (IPD).

REFERENCES:
- [Background] Marrouche NF, Brachmann J; CASTLE-AF Steering Committee. Catheter ablation versus standard conventional treatment in patients with left ventricular dysfunction and atrial fibrillation (CASTLE-AF) - study design. Pacing Clin Electrophysiol. 2009 Aug;32(8):987-94. doi: 10.1111/j.1540-8159.2009.02428.x. PMID 19659616
- [Derived] Brachmann J, Sohns C, Andresen D, Siebels J, Sehner S, Boersma L, Merkely B, Pokushalov E, Sanders P, Schunkert H, Bansch D, Dagher L, Zhao Y, Mahnkopf C, Wegscheider K, Marrouche NF. Atrial Fibrillation Burden and Clinical Outcomes in Heart Failure: The CASTLE-AF Trial. JACC Clin Electrophysiol. 2021 May;7(5):594-603. doi: 10.1016/j.jacep.2020.11.021. Epub 2021 Feb 24. PMID 33640355
- [Derived] Marrouche NF, Brachmann J, Andresen D, Siebels J, Boersma L, Jordaens L, Merkely B, Pokushalov E, Sanders P, Proff J, Schunkert H, Christ H, Vogt J, Bansch D; CASTLE-AF Investigators. Catheter Ablation for Atrial Fibrillation with Heart Failure. N Engl J Med. 2018 Feb 1;378(5):417-427. doi: 10.1056/NEJMoa1707855. PMID 29385358
- See also: Click here for more information about this study: CASTLE-AF — http://www.castle-af.org